CLINICAL TRIAL: NCT06181292
Title: Phase IIb/III, Double-Blind, Randomised, Active-Controlled, Multi-Center, Non-Inferiority Clinical Trial, to Assess the Safety and Immunogenicity of a Booster Vaccination with an Adapted Recombinant Protein RBD Fusion Homodimer Candidate Against SARS-CoV-2, in Adults Vaccinated Against COVID-19
Brief Title: Safety and Immunogenicity of a Booster Vaccination with an Adapted Vaccine
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hipra Scientific, S.L.U (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HIPRA-HH-14
Record Dates: First submitted 2023-11-28; First posted 2023-12-26 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: SARS-CoV2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PHH-1V81 (Experimental): One dose of 40ug of PHH-1V81, administered intramuscularly
  Interventions: Biological: PHH-1V81
- Comirnaty Omicron XBB1.5 (Active Comparator): One dose of 30ug of Comirnaty Omicron XBB1.5, administered intramuscularly
  Interventions: Biological: Comirnaty Omicron XBB1.5

INTERVENTIONS:
Biological: PHH-1V81 — booster of PHH-1V81
  Arms: PHH-1V81
Biological: Comirnaty Omicron XBB1.5 — booster of Comirnaty Omicron XBB1.5
  Arms: Comirnaty Omicron XBB1.5

SUMMARY:
This is a phase IIb/III, double-blind, randomised, active-controlled, multi-centre, non-inferiority clinical trial that aims to determine safety, tolerability and immunogenicity of a booster vaccination with a recombinant protein receptor binding domain (RBD) fusion homodimer of XBB.1.16 adapted candidate against SARS-CoV-2 developed by HIPRA (PHH-1V81).

DETAILED DESCRIPTION:
This is a phase IIb/III, double-blind, randomised, active-controlled, multi-centre, non-inferiority clinical trial that aims to determine safety, tolerability and immunogenicity of a booster vaccination with a recombinant protein receptor binding domain (RBD) fusion homodimer of XBB.1.16 adapted candidate against SARS-CoV-2 developed by HIPRA (PHH-1V81).

Approximately 612 participants who have received a primary scheme with an EU-approved mRNA vaccine (two doses) and at least one booster dose of an EU-approved mRNA vaccine against COVID-19, will be randomly assigned to the following two treatment arms in a PHH-1V81 : Comirnaty (Omicron XBB.1.5) 2:1 ratio:

* PHH-1V81 vaccine arm: Approximately 408 adults will receive a booster dose of PHH-1V81 (HIPRA adapted vaccine).
* Comirnaty vaccine arm: Approximately 204 adults will receive a booster dose of Comirnaty Omicron XBB.1.5.

Participants will be stratified before randomisation by age group (approximately 10% of adults ≥60 years old), and by number of doses previously received.

All participants will receive a booster dose of PHH-1V81 or Comirnaty Omicron XBB.1.5 at Day 0 and will be followed for 6 months. All subjects will be closely observed for 15 minutes after vaccination on site.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 or older at Day 0
* Are willing and able to sign the informed consent and can comply with all study visits and procedures
* Participant must have received a primary scheme of an EU-approved mRNA vaccine (2 doses) and at least one booster dose with an EU-approved mRNA vaccine. Last booster dose must have been administered at least 6 months before Day 0.
* Having a negative Rapid Antigen Test for COVID-19 at Day 0 prior to vaccination.
* Adults determined by clinical assessment, including medical history and clinical judgement, to be eligible for the study, including adults with pre-existing chronic and stable diseases (non-immunocompromised), if these are stable and well-controlled according to the investigator's judgment.
* Uses an accepted method of contraception

Exclusion Criteria:

* Participant with an acute illness with fever ≥ 38.0°C at Day 0 or within 24 hours prior to vaccination. Afebrile participants with minor illnesses can be enrolled at the discretion of the investigator
* Participant with a medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behaviour that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Participant with history of severe adverse reaction associated with a vaccine and/or severe allergic reaction (e.g. anaphylaxis) to any component of the study intervention
* Immunocompromised individuals defined as those with primary and secondary immune deficiencies and those receiving chemotherapy or immunosuppressant drugs other than steroids and glucocorticoids (maximum 30mg/day of prednisone, or equivalent, by any administration route for a maximum of 30 consecutive days), within 90 days prior to vaccination
* Participant with a bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection
* Have receipt of blood-derived immune globulins, blood, or blood-derived products in the past 3 months
* Participation in other studies involving study intervention if last dose is within 28 days prior to screening and/or it is planned to receive during study participation
* Received any non-study vaccine within 14 days before or after screening. For live or attenuated vaccines, 4 weeks before or after screening
* Received any COVID-19 vaccines other than EU-approved mRNA vaccines
* Received any Omicron XBB adapted vaccine before Day 0
* COVID-19 infection diagnosed in the previous 6 months before Day 0. History of COVID-19 infections is allowed
* History of a diagnosis or other conditions that, in the judgment of the investigator, may affect study endpoint assessment or compromise participant safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 913 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
Number, percentage and characteristics of solicited local and systemic AEs, unsolicited AEs, SAEs, AESIs and MAAEs | 0, 7, 14, 91 and 182 days post-vaccination
  To assess the safety and tolerability of a PHH-1V81 booster in adults who previously received primary vaccination and at least one booster dose of an EU-approved mRNA vaccine
Neutralising antibody titers of PHH-1V81 booster at Day 0 and 14 | 0 and 14 days post-vaccination
  To determine and compare the changes in immunogenicity measured by pseudovirus neutralisation assay (PBNA) against Omicron XBB.1.16 variant at Baseline and Day 14 in the PHH-1V81 vaccine arm versus the Comirnaty arm.

SECONDARY OUTCOMES:
Neutralising antibody titers of PHH-1V81 booster at Day 91 and 182 | 91 and 182 days post-vaccination
  To determine and compare the changes in immunogenicity measured by PBNA against Wuhan, Omicron BA.1 and Omicron XBB.1.5 at Baseline and at Days 14, 91 and 182, and Omicron XBB.1.16 at Days 91 and 182, after vaccination in the PHH-1V81 vaccine arm vs. the Comirnaty arm.
Total binding antibody titers of PHH-1V81 booster at Days 0, 14, 91 and 182 | 0, 14, 91 and 182 days post-vaccination
  To evaluate and compare the immunogenicity measured by means of total antibody against Receptor Binding Domain of the Spike protein of SARS-CoV-2, measured by an electrochemiluminescence immunoassay (ECLIA) at Baseline and at Days 14, 91 and 182 in the PHH-1V81 vaccine arm vs the Comirnaty arm.

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Prat, Study Director — Hipra Scientific, S.L.U
Locations (10):
- Spain (10):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital HM Delfos, Barcelona, Barcelona
  - CAP Centelles, Centelles, Barcelona
  - Hospital Josep Trueta, Girona, Girona
  - Hospital HM Sanchinarro, Madrid, Madrid
  - Hospital Quironsalud Madrid, Madrid, Madrid
  - Hospital HM Puerta del Sur, Móstoles, Madrid
  - Hospital Regional de Málaga, Málaga, Málaga
  - Hospital Clínico Universitario de Valencia, Valencia, Valencia
  - Hospital de Cruces, Barakaldo, VIZCAYA

IPD SHARING:
Plan to Share IPD: No